CLINICAL TRIAL: NCT00495183
Title: Efficacy of Caffeine, With and Without Biperiden, as a Maintenance Treatment for Cocaine Dependence
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Miguel Casas Brugué, Servei de Psiquiatria. Hospital Universitari Vall d'Hebron
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAF-MT; eudraCT 2005-06-01
Record Dates: First submitted 2007-06-29; First posted 2007-07-02 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-05

CONDITIONS: Cocaine Dependence
Keywords: cocaine dependence; cocaine use; CNS stimulants; caffeine; biperiden; placebo
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Caffeine; Biperiden

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): caffeine + placebo
  Interventions: Drug: caffeine
- 2 (Experimental): caffeine + biperiden
  Interventions: Drug: caffeine; Drug: Biperiden
- 3 (Placebo Comparator): Placebo+placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: caffeine — caffeine from 300 to 1200 mg/d or 15 mg/kg/d, divided in 3 doses per day.
  Other Names: Durvitan
  Arms: 1; 2
Drug: Biperiden — Biperiden 2-4 mg/d, divided in 2 doses per day.
  Other Names: Akineton
  Arms: 2
Drug: Placebo — Placebo
  Arms: 3

SUMMARY:
The aim of this study is to assess the efficacy of caffeine compared to placebo as a maintenance treatment for cocaine dependence. Caffeine potentiation with biperiden will be also studied.

Ninety patients with snorted/sniffed cocaine dependence will be randomized to receive caffeine (300 - 1200 mg t.i.d.) plus biperidene (8 mg b.i.d.) caffeine (300 - 1200 mg t.i.d.) with placebo or placebo during 10 days in an in-hospital setting.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of cocaine dependence, according to DSM-IV-TR criteria
* age between 18 and 60 years
* current cocaine use, confirmed by a positive urine drug screen for cocaine the week prior to admission.
* demonstrated capacity to grant informed consent and sign the pertinent informed consent form.
* place of residence compatible with attendance at the center.
* for women, willingness to use effective contraceptive measures during the study.

Exclusion Criteria:

* diagnosis of a severe medical disorder that could interfere with the study
* presence of an organic pathology for which methylxanthines or biperidene administration is contraindicated
* serum liver transaminase levels 3 times higher than normal values
* pregnancy and breast-feeding
* neuroleptic medication treatment in the past 6 weeks
* current treatment, or anticipation that the patient may need to initiate treatment during the study, with drugs that may interact with study medication.
* current diagnosis of a major mental disorder.
* awareness of a situation that could prevent the patient's participation in the study (e.g. serving a sentence)
* current participation in another research project.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-07 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
survival | 22 weeks
cocaine use | 22 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Miquel Casas, Prof., Principal Investigator — Hospital Universitari Vall d'Hebron Barcelona, Catalonia, Spain
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Catalonia, Spain